CLINICAL TRIAL: NCT04900610
Title: Vitamin K In PEritonial DIAlysis (VIKIPEDIA)
Brief Title: The Effect of Vitamin K2 Supplementation on Arterial Stifness and Cardiovascular Events in PEritonial DIAlysis
Acronym: VIKIPEDIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Nattopharma ASA (Industry)
Responsible Party: Principal Investigator, Vaios Vasileios, Principal Investigator, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 235/14.05.2021
Record Dates: First submitted 2021-05-19; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Vitamin K Deficiency; End Stage Renal Disease; Peritoneal Dialysis; Arterial Stiffness; Cardiovascular Morbidity; Mortality
Keywords: Vitamin K; Menaquinone-7; Peritoneal dialysis; Arterial stifness; Cardiovascular; Chronic Kidney Disease; End Stage Renal Disease
MeSH Terms: conditions — Vitamin K Deficiency; Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Multi-centre, placebo-controlled, randomized, open-label intervention clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin K2 (Active Comparator): 1mg/day per os
  Interventions: Dietary Supplement: MenaQ7 ®, Nattopharma, ASA, Hovik, Norway
- Placebo (Placebo Comparator): matching placebo
  Interventions: Dietary Supplement: MenaQ7 ®, Nattopharma, ASA, Hovik, Norway

INTERVENTIONS:
Dietary Supplement: MenaQ7 ®, Nattopharma, ASA, Hovik, Norway — daily per os supplementation of 1mg MK-7

SUMMARY:
VIKIPEDIA is a multi-centre, placebo-controlled, randomized, open-label intervention clinical trial on Peritoneal Dialysis (PD) patients. At baseline the investigators will recruit End-Stage Renal Disease patients undergoing PD and randomize them to either daily per os supplementation of 1mg menaquinone-7 or placebo for 1.5 year. The investigators will study the effect of vitamin K2 supplementation (through normalization of dp-ucMGP) on arterial stifness and the occurence of cardiovascular events. The investigators will also cosider as secondary endpoints, mortality, central aortic blood pressure and indices of 24h-ambulatory blood pressure.

DETAILED DESCRIPTION:
VIKIPEDIA is a multi-centre, placebo-controlled, randomized, open-label intervention clinical trial on PD patients. The study protocol was developed in accordance with the Helsinki Declaration of Human Rights and the Good Clinical Practice Guidelines and Standard Protocol Items: Recommendations for Intervention Trials, was approved by the Ethics Committee/Scientific Council of the Medical School of Aristotle University of Thessaloniki (235/14.05.2021) All participants will provide a structured, written, informed consent. Three university, tertiary hospitals in Northern Greece with major, referral PD units will participate in the study. The patients will be recruited within 1 year. At baseline, all eligible patients who have provided a written, informed consent will be enrolled in the study. Αortic stiffness and vitamin K status will be assessed by PWV and plasma dp-ucMGP levels respectively. Before randomization, the investigators will draw blood (serum and plasma) and PD fluid samples from all patients to measure blood count and routine biochemical parameters, including urea, creatinine, potassium, sodium, calcium, phosphorus, c-reactive protein, alkaline phosphatase, albumin, parathormone, 25-OH D3, magnesium, glycated hemoglobin, thyroid function hormones. Since both vitamin D and magnesium are considered of utmost importance in vitamin K metabolism, after baseline, patients with vitamin D and/or magnesium depletion will be treated with oral supplements to achieve normal levels of both elements, before randomization. The cohort will then be categorized to one of the two groups (placebo or active group) and the treatment period will last 1.5 years. To ensure that the two parallel groups will include patients that will not differ significantly in vitamin K and stiffness, patients will be accordingly stratified. After randomization, all patients will continue their routine, standard medical treatment and patients in the treatment group will additionally receive daily, per os 1 mg of vitamin K2 (MenaQ7 ®, Nattopharma, ASA, Hovik, Norway).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* At least 3 months on PD
* Life expectancy of ≥ 18 months

Exclusion Criteria:

* Liver disease
* Drug or alcohol abuse
* Pregnancy or breast-feeding
* Treatment with phosphate binders (sevelamer)
* Ongoing malignancy or severe inflammatory disease diagnosis
* Use of vitamin K antagonist or vitamin K supplements during the past 3 months
* Diagnosis of severe gut-disease (inflammatory or short bowel disease) or gastrointestinal malabsorption
* Mental disorder rendering the patient unable to conform with the instructions and fully understand the nature, aim and possible side-effects of the supplementation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Progression of arterial stifness | 1.5 years
  Change in pulse wave velocity
Non fatal cardiovascular events | 1.5 years
  Number of patients presenting acute myocardial infarction, acute coronary syndrome, embolism, peripheral arterial disease and stroke

SECONDARY OUTCOMES:
Mortality | 1.5 years
  Number of participants who willl die from any cause
PD adequacy | 1.5 years
  Number of patients with preserved residual renal function
PD clearance | 1.5 years
  Change in Kt/V
Infections/peritonitis | 1.5 years
  Rate of infections and peritonitis
Parathormone homeostasis | 1.5 year
  Changes in serum parathormone
Calcium phosphorus homeostasis | 1.5 year
  Changes in the calcium phosphorus product
Fractures | 1.5 years
  Incidence of fractures
Joint/muscle pain | 1.5 years
  Incidence of pain in muscles and/or joints
24-hour ambulatory BP/aortic systolic BP | 1.5 years
  Change in indices of ambulatory BP and aortic systolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Stefanos Roumeliotis, MD, PhD, Principal Investigator — 1st Department of Internal Medicine, Medical School, Aristotle University of Thessaloniki; Vassilios Liakopoulos, Professor, Principal Investigator — 1st Department of Internal Medicine, Medical School, Aristotle University of Thessaloniki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Roumeliotis S, Roumeliotis A, Dounousi E, Eleftheriadis T, Liakopoulos V. Vitamin K for the Treatment of Cardiovascular Disease in End-Stage Renal Disease Patients: Is there Hope? Curr Vasc Pharmacol. 2021;19(1):77-90. doi: 10.2174/1570161118666200320111745. PMID 32196451
- [Result] Roumeliotis S, Dounousi E, Eleftheriadis T, Liakopoulos V. Association of the Inactive Circulating Matrix Gla Protein with Vitamin K Intake, Calcification, Mortality, and Cardiovascular Disease: A Review. Int J Mol Sci. 2019 Feb 1;20(3):628. doi: 10.3390/ijms20030628. PMID 30717170
- [Result] Roumeliotis S, Dounousi E, Salmas M, Eleftheriadis T, Liakopoulos V. Vascular Calcification in Chronic Kidney Disease: The Role of Vitamin K- Dependent Matrix Gla Protein. Front Med (Lausanne). 2020 Apr 24;7:154. doi: 10.3389/fmed.2020.00154. eCollection 2020. PMID 32391368
- [Result] Xu Q, Guo H, Cao S, Zhou Q, Chen J, Su M, Chen S, Jiang S, Shi X, Wen Y. Associations of vitamin K status with mortality and cardiovascular events in peritoneal dialysis patients. Int Urol Nephrol. 2019 Mar;51(3):527-534. doi: 10.1007/s11255-019-02080-x. Epub 2019 Jan 28. PMID 30689181
- [Result] Peeters FECM, van Mourik MJW, Meex SJR, Bucerius J, Schalla SM, Gerretsen SC, Mihl C, Dweck MR, Schurgers LJ, Wildberger JE, Crijns HJGM, Kietselaer BLJH. Bicuspid Aortic Valve Stenosis and the Effect of Vitamin K2 on Calcification Using 18F-Sodium Fluoride Positron Emission Tomography/Magnetic Resonance: The BASIK2 Rationale and Trial Design. Nutrients. 2018 Mar 21;10(4):386. doi: 10.3390/nu10040386. PMID 29561783
- [Result] Haroon SW, Tai BC, Ling LH, Teo L, Davenport A, Schurgers L, Teo BW, Khatri P, Ong CC, Low S, Yeo XE, Tan JN, Subramanian S, Chua HR, Tan SY, Wong WK, Lau TW. Treatment to reduce vascular calcification in hemodialysis patients using vitamin K (Trevasc-HDK): A study protocol for a randomized controlled trial. Medicine (Baltimore). 2020 Sep 4;99(36):e21906. doi: 10.1097/MD.0000000000021906. PMID 32899022
- [Result] Vaios V, Georgianos PI, Vareta G, Dounousi E, Dimitriadis C, Eleftheriadis T, Papagianni A, Zebekakis PE, Liakopoulos V. Clinic and Home Blood Pressure Monitoring for the Detection of Ambulatory Hypertension Among Patients on Peritoneal Dialysis. Hypertension. 2019 Oct;74(4):998-1004. doi: 10.1161/HYPERTENSIONAHA.119.13443. Epub 2019 Aug 12. PMID 31401878
- [Derived] Roumeliotis S, Roumeliotis A, Georgianos PI, Thodis E, Schurgers LJ, Maresz K, Eleftheriadis T, Dounousi E, Tripepi G, Mallamaci F, Liakopoulos V. VItamin K In PEritonial DIAlysis (VIKIPEDIA): Rationale and study protocol for a randomized controlled trial. PLoS One. 2022 Aug 17;17(8):e0273102. doi: 10.1371/journal.pone.0273102. eCollection 2022. PMID 35976944